CLINICAL TRIAL: NCT05622214
Title: An Open Label, Pilot Study Assessing the Efficacy and Tolerability of 12-weeks Treatment With Almond and Buckwheat Based Formula in Pediatric Patients With Active Eosinophilic Esophagitis (EoE)
Brief Title: The Efficacy and Tolerability of 12-weeks Treatment With Almond and Buckwheat Based Formula in Pediatric Patients With Active EoE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Else Nutrition GH Ltd (Industry)
Responsible Party: Principal Investigator, Ron Shaoul MD, Director, Pediatric Gastroenterology institute, Rambam Health Care Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0400-21-RMB
Record Dates: First submitted 2022-11-14; First posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Plant based nutrition (Experimental): Plant based nutritional formula based on almond and buckwheat
  Interventions: Dietary Supplement: Else nutrition formula

INTERVENTIONS:
Dietary Supplement: Else nutrition formula — Plant based nutrition from almond and buckwheat

SUMMARY:
Eosinophilic esophagitis (EoE) is a chronic, relapsing, immune-mediated esophageal disease. Clinical manifestations in infants and toddlers generally include vomiting, food refusal, choking with meals and, less commonly, failure to thrive. The management of the disease includes dietary and pharmaceutical interventions, and the goal of the treatment should ideally be both the resolution of symptoms and the normalization of the macroscopic and microscopic abnormalities. Milk is the most common food trigger identified, followed by wheat, soy, and eggs. The aim of the study is to examine the tolerability of a new plant based formula made of minimally processed almond and buckwheat and enriched with vitamins and minerals.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with active EoE (naïve and experienced)
* Ages 1-18 years

Exclusion Criteria:

* Change in dosing of Proton pump inhibitors (PPI) medication
* Local steroid treatment < 1 month
* Refusal to comply with study protocol
* Known allergy to almonds and buckwheat
* Use of dairy during the study

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-07-24 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in Pediatric Eosinophilic Esophagitis Symptom Severity Module (PEESS), endoscopic and histological scoring | 12 weeks
  Improvement in PEESS, endoscopic and histological scoring (assessed at week 0 and week 12)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Shaoul, Dr., Principal Investigator — Rambam Health Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel